CLINICAL TRIAL: NCT04142372
Title: Tissue Microarray of Hematological Malignancies: Search for Novel Regulators of Disease Pathology Across Disease Entities
Brief Title: Tissue Microarray of Hematological Malignancies
Acronym: HemaTMA
Status: Active, not recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); University of Eastern Finland (Other); Fimlab Oy (Unknown); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Matti Vänskä, Principal Investigator, MD PhD, Tampere University
Other Study IDs: R19060B
Record Dates: First submitted 2019-09-18; First posted 2019-10-29 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Hematological Malignancies
Keywords: leukemia; lymphoma; biomarker; prognosis; myeloma; myelodysplasia; myeloproliferative disorder; diagnostics; tissue microarray; proteomics; genomics; clinical outcome; biobanking; digitalization; data mining; hematology; oncology; pathology; bioinformatics; real world data; hematological malignancy; survival; treatment response
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Neoplasms, Plasma Cell; Anemia, Refractory, with Excess of Blasts; Myeloproliferative Disorders; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Diagnostic samples containing cells and tissues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to create new tools for improving management of patients with hematological malignancies by combining extensive clinical data from patients newly diagnosed with hematological malignancies and innovative laboratory analyses made on available tissue samples in regional biobanks from these patients.

DETAILED DESCRIPTION:
Firstly, clinical information is collected on all hematological malignancies diagnosed in our hospital district area retrospectively between the years 2000 and 2019. Clinical outcomes, laboratory results, clinically relevant diagnoses, characteristics defining clinical stage and established prognostic parameters are gathered.

Simultaneously a tissue microarray (TMA) of diagnostic samples is compiled using representative annotated tissue areas. This TMA is used in combination with additional control material to identify prognostic and predictive biomarkers.

A combined microarray dataset of hematological malignancies (Hemap) is utilized to point out genes of possible drug targets, disease specific markers, prognostic markers, or predictive markers.

The clinical datasets and Hemap dataset is ultimately utilized to gain knowledge, new tools for prognostication and diagnostics, and targets for treatment. Artificial intelligence -assisted differential diagnostics will be tested.

ELIGIBILITY:
Inclusion Criteria:

* hematological malignancy/neoplasm

Exclusion Criteria:

* Non-sufficient data available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with new hematological malignancies 1.1.2000- 30.4.2019
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the first line treatment up to the end of the study period (April 2019).
  Time from the first line treatment for hematological malignancy until the date of first documented relapse or transformation or death of any cause, whichever came first, assessed up to the end of the study period (April 2019).
Overall survival (OS) | From the diagnosis up to the end of the study period (April 2019).
  Survival time from the diagnosis of hematological malignancy until the date of death of any cause, assessed up to the end of the study period (April 2019).
Response to treatment | From the first line treatment up to the end of the study period (April 2019).
  Best response to the first line treatment for the hematological malignancy, according to malignancy in question, e.g. complete response (CR), stringent complete response (sCR), partial response (PR), very good partial response (VGPR), stable disease (SD), progressive disease (PD), treatment failure, clinical response, hematological response etc.
Event-free survival (EFS) | From the first line treatment up to the end of the study period (April 2019).
  Survival time from the first line treatment for hematological malignancy until any primary event (death, relapse, disease progression/transformation, secondary malignancy, resistant disease etc.), whichever came first, assessed up to the end of the study period (April 2019).

SECONDARY OUTCOMES:
Sepsis or other life-threatening infection | From the first line treatment up to the end of the study period (April 2019).
  Fulminant infection after diagnosis
Multiple organ failure | From the first line treatment up to the end of the study period (April 2019).
  Altered organ function in acutely ill patient
Thrombo-embolism | From the first line treatment up to the end of the study period (April 2019).
  Venous thromboembolism
Disease transformation | From the diagnosis up to the end of the study period (April 2019).
  Hematological malignancy transforms into another malignancy
ICU admission | From the first line treatment up to the end of the study period (April 2019).
  Admission to intensive care unit
Adverse effects | From the first line treatment up to the end of the study period (April 2019).
  Treatment-related adverse effects/events
Secondary malignancy | From the first line treatment up to the end of the study period (April 2019).
  Secondary malignancy after the diagnosis of hematological malignancy
Relapse | From the first line treatment up to the end of the study period (April 2019).
  Relapse after or during the treatment.
Complete remission | From the first line treatment up to the end of the study period (April 2019).
  Complete remission after the treatment
Time to complete remission | From the first line treatment up to the end of the study period (April 2019).
  Time to complete remission
Best response | From the first line treatment up to the end of the study period (April 2019).
  Best response e.g. hematological remission, molecular remission, radiological remission
Time to best response | From the first line treatment up to the end of the study period (April 2019).
  Time to best response e.g. hematological remission, molecular remission, radiological remission

CONTACTS AND LOCATIONS:
Overall Officials: Artturi Mäkinen, MD, Principal Investigator — Tampere University; Olli Lohi, MD, PhD, Study Chair — Tampere University; Merja Heinäniemi, PhD, Study Chair — University of Eastern Finland; Matti Vänskä, MD, PhD, Principal Investigator — Tampere University Hospital; Tiina Lyly-Yrjänäinen, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere Univerisity Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided